CLINICAL TRIAL: NCT02210195
Title: Pharmacological Treatment of Comorbid Alcohol and Marijuana Withdrawal and Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, Principal Investigator, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA030988-04S1; R01DA030988-04S1 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-06 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Cannabis Dependence; Alcohol Dependence; Cannabis Use Disorder; Alcohol Use Disorder
Keywords: Cannabis Treatment; Alcohol Treatment; Alcohol-Related Disorders; Cannabis-Related Disorders; Substance-Related Disorders; Emend; NK1 receptor antagonist; Alcohol; Cannabis; aprepitant
MeSH Terms: conditions — Marijuana Abuse; Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: aprepitant 125 mg/day (Active Comparator): 125 mg aprepitant daily for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
  Interventions: Drug: aprepitant; Behavioral: Manual-guided behavioral counseling
- Placebo 125mg/d (Placebo Comparator): Matched placebo pill given daily for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
  Interventions: Drug: Placebo; Behavioral: Manual-guided behavioral counseling

INTERVENTIONS:
Drug: aprepitant — 125 mg daily for 8 weeks.
  Other Names: Emend
  Arms: Experimental: aprepitant 125 mg/day
Drug: Placebo — Placebo daily for 8 weeks.
  Arms: Placebo 125mg/d
Behavioral: Manual-guided behavioral counseling — Standardized manual-guided behavioral counseling performed 1 time per week for 8 weeks in conjunction with study drug or placebo.
  Other Names: Manual-guided therapy

SUMMARY:
The primary aim of the supplemental study is to provide POC testing of aprepitant as a treatment for comorbid alcohol and cannabis dependence. The data analysis plan specified in the parent grant will likewise be applied to the supplemental project to test for effects of aprepitant vs placebo on measures of alcohol and cannabis use and protracted withdrawal. The primary hypothesis is that subjects treated with aprepitant will have significantly less alcohol and marijuana use than subjects treated with placebo.

DETAILED DESCRIPTION:
Consistent with the scope and methods of the parent grant, this was a randomized, double-blind, placebo-controlled, parallel groups, Phase II, single-site, 8-week clinical trial of aprepitant 125 mg/d or placebo. Participants were 20 outpatients seeking treatment for concurrent alcohol and cannabis dependence. All participants received weekly protocol-specific counseling. Research assessments occurred weekly through the treatment phase of the 8-week study. Post treatment follow-up assessments occurred at Weeks 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 18-70 years of age
* Meets DSM IV criteria for current alcohol and cannabis dependence
* Seeking research-based outpatient treatment for alcohol and cannabis dependence that involves daily oral medication
* Negative BAC and a CIWA score < 9 at randomization

Exclusion Criteria:

* Significant medical disorders or use of medications that will increase potential risk or influence study outcomes
* Females who are pregnant, nursing or who are sexually active with child-bearing potential and refuse to use an effective, non hormonal method of birth control during the study and for up to 4 weeks after study termination• Treatment with an investigational drug during the previous month
* Prior treatment with NK1 antagonists
* Participants for whom treatment is being mandated by a legal authority• Inability to understand and/or comply with the provisions of the protocol and consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant: 125mg/Day: 125mg/d aprepitant for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
- Matched Placebo: Matched Placebo daily for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
Period: Overall Study
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Started | 10 | 10
Completed | 6 | 10
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (13.5) | 35.5 (9.3) | 35.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 in Cannabis Use Using Urinary CN-THCCOOH Levels at Week 8
Description: Urinary THC/Cr ratio, also known as CN-THCCOOH (creatinine normalized tetrahydrocannabinol carboxylic acid), is a highly sensitive and specific quantitative analytic procedure to determine current marijuana metabolite levels in the urine as well as new marijuana use or abstinence. Gas chromatography mass spectrometric levels of 11-nor-9-carboxy-9-THC (THC-COOH), the primary marijuana metabolite, are normalized to the urine creatinine (CN) concentration to reduce the variability of drug measurement attributable to urine dilution. Negative values indicate decreased use. Change = (Week 8 value - Week 0 value).
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Number analyzed (Participants) | 6 | 10
ng/mg | 198.3 (389.4) | 55.9 (239.3)

2. Primary Outcome: Change From Week 0 in Drinking Quantity and Frequency Using Drinks Per Week at Week 8
Description: Standard drinks are equivalent to 14 grams of pure alcohol and number of drinks are assessed with Timeline Follow-Back (TLFB) methods. Change = (Week 8 - Week 0). More negative values indicate less use of alcohol.
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Number analyzed (Participants) | 6 | 10
drinks/week | -21.0 (16.1) | -10.7 (17.1)

ADVERSE EVENTS:
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant: 125mg/Day (N=10) | Matched Placebo (N=10)
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No